CLINICAL TRIAL: NCT07322874
Title: The Effect of Menstrual Cycle on Exercise-induced Muscle Damage
Brief Title: Menstrual Cycle and Exercise-induced Muscle Damage
Acronym: MC-EIMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chariklia K. Deli (Other)
Responsible Party: Sponsor-Investigator, Chariklia K. Deli, Associate Professor, University of Thessaly
Organization: University of Thessaly (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: Menstrual Cycle - EIMD
Record Dates: First submitted 2025-12-07; First posted 2026-01-07 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Menstrual Cycle Phase
Keywords: menstrual cycle; follicular phase; luteal phase; exercise-induced muscle damage; muscle performance; muscle soreness
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Follicular phase (Experimental): The participants will perform downhill running (-15% slope) on a treadmill at 70% of HRmax followed by running on a horizontal level (0% slope) at 95% HRmax until exhaustion, during the follicular phase
  Interventions: Other: Exercise during follicular phase
- Luteal phase (Experimental): The participants will perform downhill running (-15% slope) on a treadmill at 70% of HRmax followed by running on a horizontal level (0% slope) at 95% HRmax until exhaustion, during the luteal phase
  Interventions: Other: Exercise during luteal phase

INTERVENTIONS:
Other: Exercise during follicular phase — The participants will perform downhill running (-15% slope) on a treadmill at 70% of HRmax followed by running on a horizontal level (0% slope) at 95% HRmax until exhaustion, during the follicular phase
  Arms: Follicular phase
Other: Exercise during luteal phase — The participants will perform downhill running (-15% slope) on a treadmill at 70% of HRmax followed by running on a horizontal level (0% slope) at 95% HRmax until exhaustion, during the luteal phase
  Arms: Luteal phase

SUMMARY:
The aim of the study is to investigate the effect of the different menstrual cycle phases on the recovery from exercise-induced muscle injury in eumenorrheic women. For this purpose, in a cross-over, randomized study, at least 10 healthy eumenorrheic women aged 18-35 years will participate. In a random order, the participants will perform 45 min downhill (-15% slope) running on a treadmill at 70% HRmax followed by a maximal time-trial (95% HRmax) to exhaustion: i) during the follicular phase and ii) during the luteal phase. Before the exercise protocol, as well as at 24 h, 48 h and 72 h following exercise, complete blood count, delayed onset of muscle soreness (DOMS), creatine kinase activity, countermovement jump, isometric, concentric and eccentric strength of knee extensors and knee flexors, will be assessed. In addition, lactic acid concentration will be assessed before and immediately following exercise, and DOMS will be assessed immediately after the end of exercise. Following a washout period of ≥28 days (depending on the length of the menstrual cycle), participants will repeat the exact same procedure for the remaining phase of the menstrual cycle.

DETAILED DESCRIPTION:
Research in the field of athletic training and rehabilitation, has traditionally focused on men, ignoring the physiological differences between sexes that may significantly affect athletic performance and recovery following exercise-induced muscle damage (EIMD). According to recent reviews of research in sports and exercise medicine, female representation is particularly limited, with only 4% - 13% of studies including women [1]. However, the number of females' participation in regular exercise and sports constantly increases, therefore it is imperative to define EIMD in women.

Except for being limited, most of the existing studies in women have been conducted during the early follicular phase of the cycle, when estrogen and progesterone levels are low, so that women's hormonal profile resembles that of men [2], in order to avoid any fluctuations [3]. However, this approach limits our understanding of the effects of the other phases of the cycle, such as the luteal phase, on performance and exercise-induced inflammation, and thus on women's ability to train and perform.

Although limited, some data suggest the influence of different phases of the menstrual cycle on both performance and exercise-induced muscle injury. For example, women's thermoregulatory levels are higher during the luteal phase of the cycle, which may affect their cardiovascular performance and endurance [4]. Similar data suggest that hormonal fluctuations may also affect recovery from EIMD [5]. Indicatively, the concentration of CK and IL-6 24 h and 72 h following 90 min of continuous running at 70% of VO2max was higher during the follicular phase [6].

Considering the above, research regarding the effect of the different phases of the menstrual cycle on performance and EIMD, it is crucial for the effective design of individualized training programs depending on the phase of the menstrual cycle, to improve performance and avoid injuries in women.

The aim of the study is to investigate the effect of the different menstrual cycle phases on the recovery from EIMD in eumenorrheic women.

According to an initial power analysis performed (probability error: 0.05, power: 0.80), a number of 8-10 individuals is required in order to identify statistically significant differences. Therefore, at least 10 participants will be included in the present study.

The design of the present study is cross-over, randomized and will be conducted in two cycles. The participants, after being informed about the study, as well as the benefits and potential risks, will sign an informed consent for participation in the study. Before the initiation of the data collection, familiarization of the participants with the assessment tests and the exercise protocol at low intensity, will precede. Also, the participants will provide a 7-days diet recall before their participation in the first experimental condition. Subsequently, baseline measurements will be performed at the Biochemistry, Physiology and Exercise Nutrition Laboratory (SmArT Lab), Department of Physical Education and Sports, University of Thessaly: anthropometric characteristics (body height, body mass, body mass index), body composition (body fat percentage, lean body mass, fat mass, bone density), aerobic capacity (VO2max). Subsequently, in a random order, the participants will perform 45 min of submaximal (at 70% HRmax) downhill (-15%) running on a treadmill followed by a maximal (95% HRmax) time-trial to exhaustion: i) during the follicular phase and ii) during the luteal phase. The randomization of the menstrual cycle phases will be done by a random integer sets generator, available online (Random.org). Before the exercise protocol, as well as 24 h, 48 h and 72 h following exercise, complete blood count (CBC), exercise-induced muscle injury [delayed onset muscle soreness (DOMS), creatine kinase (CK) activity] and muscle performance [(countermovement jump (CMJ), isometric, concentric and eccentric strength of knee extensors and knee flexors)] will be assessed. In addition, metabolism (lactic acid) will be assessed before and immediately following exercise, and DOMS will be assessed immediately after the end of exercise. Following a washout period of ≥28 days (depending on the length of the menstrual cycle), participants will repeat the exact same procedure for the remaining phase of the menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* Physically active subjects (VO2max ≥35ml/kg/min)
* Absence of musculoskeletal injury (≥6 months)
* Abstinence from the use of ergogenic supplements (≥1 month)
* Abstinence from anti-inflammatory drugs (≥1 month)
* Abstinence from participating in exercise with eccentric content for at least 7 days before exercise
* Abstinence from alcohol and energy drinks before exercise

Exclusion Criteria:

* Recent history of musculoskeletal injury (<6 months)
* Use of ergogenic performance supplements (<1 month)
* Taking anti-inflammatory drugs (<1 month)
* Participation in exercise with eccentric content in the previous 7 days before exercise
* Consumption of alcohol and energy drinks before exercise

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Changes in Creatine kinase (CK) activity | At baseline (pre), post-, 24 hours post-, 48 hours post-, 72 hours post-trial
  CK activity will be measured in plasma using a Clinical Chemistry Analyzer with commercially available kits.
Changes in delayed onset of muscle soreness (DOMS) | At baseline (pre), post-, 24 hours post-, 48 hours post-, 72 hours post-tria
  DOMS of knee extensors, knee flexors, gluteal and gastrocnemius muscles of both lower extremities will be measured during palpation of the muscle belly and the distal region after performing three repetitions of a full squat.
Changes in blood lactate concentration | At baseline (pre), 4 minutes post-exercise
  Lactate concentration will be measured in capillary blood with a hand-portable analyzer
Changes in countermovement jump (CMJ) height | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  CMJ height will be measured with an optical system. Participants will perform 3 maximal CMJ jumps and the best effort will be recorded
Changes in isokinetic strength of knee extensors (KE) and knee flexors (KF) | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Isometric, concentric and eccentric peak torque of the KE and KF of both limbs will be assessed on an isokinetic dynamometer
Changes in complete blood count (CBC) | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  CBC (white blood cells, erythrocytes, platelets) will be measured in an hematological analyzer with commercially available reagents

SECONDARY OUTCOMES:
Differences in Estradiol concentration between trials | At late-follicular and mid-luteal phase (according to each participant's menstrual cycle length), before exercise
  Estradiol concentration will be measured in an automated analyzer with commercially available kits
Differences in Progesterone concentration between trials | At late-follicular and mid-luteal phase (according to each participant's menstrual cycle length), before exercise
  Progesterone concentration will be measured in an automated analyzer with commercially available kits
Body weight | At late-follicular and mid-luteal phase (according to each participant's menstrual cycle length), before exercise
  Body weight will be measured on a beam balance with stadiometer
Body height | At late-follicular and mid-luteal phase (according to each participant's menstrual cycle length), before exercise
  Body height will be measured on a beam balance with stadiometer
Body mass index (BMI) | At late-follicular and mid-luteal phase (according to each participant's menstrual cycle length), before exercise
  BMI will be calculated from the ratio of body mass/ body height squared
Body fat | At late-follicular and mid-luteal phase (according to each participant's menstrual cycle length), before exercise
  Body fat will be measured via bioelectrical impedance
Dietary intake | At baseline
  Dietary intake will be assessed using 7-day diet recalls

CONTACTS AND LOCATIONS:
Overall Officials: Chariklia K Deli, Associate Professor, MSc, PhD, Principal Investigator — University of Thessaly
Locations (1):
- Department of Physical Education and Sport Science, University of Thessaly, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roepstorff C, Steffensen CH, Madsen M, Stallknecht B, Kanstrup IL, Richter EA, Kiens B. Gender differences in substrate utilization during submaximal exercise in endurance-trained subjects. Am J Physiol Endocrinol Metab. 2002 Feb;282(2):E435-47. doi: 10.1152/ajpendo.00266.2001. PMID 11788377
- [Background] Romero-Parra N, Cupeiro R, Alfaro-Magallanes VM, Rael B, Rubio-Arias JA, Peinado AB, Benito PJ; IronFEMME Study Group. Exercise-Induced Muscle Damage During the Menstrual Cycle: A Systematic Review and Meta-Analysis. J Strength Cond Res. 2021 Feb 1;35(2):549-561. doi: 10.1519/JSC.0000000000003878. PMID 33201156
- [Background] Ruby BC, Coggan AR, Zderic TW. Gender differences in glucose kinetics and substrate oxidation during exercise near the lactate threshold. J Appl Physiol (1985). 2002 Mar;92(3):1125-32. doi: 10.1152/japplphysiol.00296.2001. PMID 11842049
- [Background] Oosthuyse T, Strauss JA, Hackney AC. Understanding the female athlete: molecular mechanisms underpinning menstrual phase differences in exercise metabolism. Eur J Appl Physiol. 2023 Mar;123(3):423-450. doi: 10.1007/s00421-022-05090-3. Epub 2022 Nov 19. PMID 36402915
- [Background] D'Eon TM, Sharoff C, Chipkin SR, Grow D, Ruby BC, Braun B. Regulation of exercise carbohydrate metabolism by estrogen and progesterone in women. Am J Physiol Endocrinol Metab. 2002 Nov;283(5):E1046-55. doi: 10.1152/ajpendo.00271.2002. PMID 12376334
- [Background] Ose BM, Eisenhauer J, Roepe I, Herda AA, Vopat BG, Vopat LM. Where Are All the Female Participants in Sports and Exercise Medicine Research? A Decade Later. Am J Sports Med. 2025 Jul;53(8):2022-2028. doi: 10.1177/03635465241278350. Epub 2025 Jan 9. PMID 39780766